CLINICAL TRIAL: NCT06136013
Title: Another Look to Exercise Prescription: Exercise Timing and the Circadian Clock in Individuals With Type 2 Diabetes and Those at Risk
Brief Title: Exercise Timing and the Circadian Clock in Individuals With Type 2 Diabetes and Those at Risk
Acronym: EX-TIMING
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Faculdade de Motricidade Humana (Other)
Collaborators: Fundação para a Ciência e a Tecnologia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: EX-TIMING_2023
Record Dates: First submitted 2023-07-26; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Exercise; Diabetes Mellitus Type 2; Glycemic Control; Inter-individual variability; Aging; Obesity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Motor Activity; Obesity

STUDY DESIGN:
Intervention Model Description: This project will consist of a randomized cross-over exercise intervention involving 2 groups: Group 1, individuals with T2DM; Group 2, age-matched older adults with overweight/obesity. Each study will consist of 3, 2-week blocks of 3 days per week of supervised post-prandial exercise using high-intensity interval training (HIIT). Between each training block, a 2-week washout period, where participants avoid structured exercise, will take place. This has been shown to be enough time to eliminate any exercise effects on insulin sensitivity and glycemic control.
  The cross-over groups are the following:
  1. morning HIIT.
  2. afternoon HIIT.
  3. evening HIIT.
  Each participant will serve as their own control, helping to account for the biological variability within the individual, as well as their individual chronotype, such as sleep/wake cycles. Participants will be randomly selected to a block order.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Morning HIIT 30-min following breakfast between 9:00 to 10:00 am. (Experimental): The exercise prescription will be standardized according to body weight and based on physical activity guidelines to achieve a weekly target of 10 kcal/kg. The duration of the exercise sessions will be based on the weekly target for energy expenditure, considering weight and individual VO2peak and will be updated at the beginning of each intervention block.
  Interventions: Behavioral: HIIT
- Afternoon HIIT 30-min following lunch between 2:00 to 3:00 pm. (Experimental): The exercise prescription will be standardized according to body weight and based on physical activity guidelines to achieve a weekly target of 10 kcal/kg. The duration of the exercise sessions will be based on the weekly target for energy expenditure, considering weight and individual VO2peak and will be updated at the beginning of each intervention block.
  Interventions: Behavioral: HIIT
- Evening HIIT 30-min following dinner between 7:00 to 8:00 pm. (Experimental): The exercise prescription will be standardized according to body weight and based on physical activity guidelines to achieve a weekly target of 10 kcal/kg. The duration of the exercise sessions will be based on the weekly target for energy expenditure, considering weight and individual VO2peak and will be updated at the beginning of each intervention block.
  Interventions: Behavioral: HIIT

INTERVENTIONS:
Behavioral: HIIT — 1 minute of exercise at 90% of their PPO, followed by a 1-minute rest at 40-60% of their peak power output using a cycle ergometer.

SUMMARY:
Many investigations have been done to determine the exercise that can elicit the greatest benefits on glycemic control and metabolic health, with findings suggesting that incorporation of higher intensity and longer duration of exercise prescribed may eliminate much of the "non-response" observed following exercise training. Even with the incorporation of higher intensity exercise into interventions aimed at improving glycemic control in individuals with type 2 diabetes mellitus (T2DM), the investigators and others continue to have mixed results, with not all individuals with T2DM obtaining benefits in insulin sensitivity and glycemic control to a given exercise training program.

Many of the metabolic processes involved in glucose homeostasis, such as insulin production and sensitivity, undergo daily circadian rhythms, controlled by cellular clock machinery located both centrally and peripherally (i.e. skeletal muscle). However, in adults with T2DM, these diurnal rhythms are impaired, with reduced insulin sensitivity in the morning, which is thought to contribute to the fasting hyperglycemia (i.e., "dawn phenomenon") observed in these individuals. Exercise may be a non-photic cue that can amplify or alter these metabolic rhythms. It has been suggested that skeletal muscle metabolic inflexibility in metabolic disorders such as overweight/obesity and T2DM is associated with reduced mitochondrial fatty acid oxidative capacity. It has been demonstrated that exercise can increase mitochondrial oxidative capacity by remodeling mitochondrial morphology and dynamics. It is unknown if potential differences in metabolic flexibility can be found in response to exercise at different times of the day.

Most of the experimental evidence originates from animal models with only 3 studies performed in humans with T2DM, which displayed conflicting results.

To overcome the shortcomings in the literature, the main objective of this research project is to assess the effects of performing exercise at different times of the day on glycemic control and related outcomes on the inter-individual response variability in glycemic control and related metabolic health parameters in two distinct populations: 1) individuals with T2DM on the most common mono-hyperglycemic drug therapy (i.e., metformin); and 2) age-matched sedentary overweight/obese individuals, where glycemic control is known to deteriorate, hence increasing the risk of developing insulin resistance and T2DM.

DETAILED DESCRIPTION:
To detect a predicted mean difference in 24-hour area under the curve (AUC) continuous glucose measure (CGM)-based glucose of 1.0 mmol/L with a within patient standard deviation (SD) of 0.85 mmol/L (24) considering a type I error of 5%, a power of 80%, and a 30% dropout rate, the investigators calculated a required sample size of 17 individuals for each group, making a total sample of 34 individuals (Group 1: T2DM; Group 2: age-matched overweight/obese).

Participants will be recruited through: flyers and posters in pharmacies, health centers and supermarkets; ads via national radios and television programs; and the database of the Portuguese Association for the Protection of Diabetics (APDP).

To improve exercise adherence, the following strategies will be implemented:

* Inform that participation in the study is completely voluntary and that all data will be confidential
* Inform people that they will be able to do physical exercise (guided by professionals) for free
* Inform that they will have individual follow-up by a personal trainer
* Inform that they will carry out several analyzes and exams free of charge that will contribute to the control of their health status
* Inform that they will be able to control their blood glucose levels and prevent or delay the complications of diabetes
* Inform that they will learn appropriate physical exercises to better control diabetes (Group 1), prevent diabetes (Group 2), and improve overall health (both Group 1 and 2) All study measurements will be collected at the Faculty of Human Kinetics, University of Lisbon. Body composition, cardiopulmonary exercise test (CPET), blood collection, metabolic flexibility, dietary records, and 24-hr CGM recording will be done at baseline as well as at the end of each 2-week intervention block. Physical activity assessment will be performed at baseline and during each 2-week washout period. The evaluations inherent to the project at baseline and at the end of each 2-week intervention block will take place on two different days.

ELIGIBILITY:
Inclusion Criteria (Group 1):

* previous diagnosis of T2DM
* currently taking metformin (Group 1 only);
* Adults aged 55 to 75 years
* Physically inactive people (i.e. with less than 20 minutes per day of exercise, maximum 3 days per week)

Exclusion Criteria (Group 1):

* Use of exogenous insulin and taking any other antihyperglycemic medication beyond metformin
* having major micro- or macro-vascular complications from T2DM
* History of cardiovascular incidents
* People with motor limitations (musculoskeletal or neurological) that limit the practice of physical exercise
* inability to provide informed consent

Inclusion Criteria (Group 2):

* BMI ≥25 without diagnosis of T2DM
* Adults aged 55 to 75 years
* Physically inactive people (i.e. with less than 20 minutes per day of exercise, maximum 3 days per week)

Exclusion Criteria (Group 2):

* History of cardiovascular incidents
* People with motor limitations (musculoskeletal or neurological) that limit the practice of physical exercise
* inability to provide informed consent

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2024-07 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Changes in 24-hour area under cover (AUC) glucose from baseline to 1, 2, and 3 months | 3 months
  Assess differences in 24-hour area under cover (AUC) glucose at different exercise times (i.e. morning, afternoon and evening) separately for individuals with T2DM and age-matched overweight/obese older adults.

SECONDARY OUTCOMES:
Changes in body mass index (BMI) from baseline to 1, 2, and 3 months | 3 months
  Participants will be weighed to the nearest 0.01kg wearing minimal clothes and without shoes and height will be measured to the nearest 0.1cm on a digital scale with an integrated stadiometer (Seca, Hamburg, Germany). From weight and height, BMI will be calculated as weight (kg) divided by the square of the height (m).
Changes in bone mineral density from baseline to 1, 2, and 3 months | 3 months
  Dual-energy X-ray absorptiometry (DXA) (Hologic Explorer-W, fan-beam densitometer, software QDR for Windows version 12.4, Waltham, USA) will be used to estimate bone mineral content and density. A whole-body scan will be performed and the attenuation of X-rays pulsed between 70 and 140 kV synchronously with the line frequency for each pixel of the scanned image that will be measured.
Changes in fat and lean body mass from baseline to 1, 2, and 3 months | 3 months
  Dual-energy X-ray absorptiometry (DXA) (Hologic Explorer-W, fan-beam densitometer, software QDR for Windows version 12.4, Waltham, USA) will be used to estimate total and regional fat mass and lean body mass.
Changes in resting metabolic rate (RMR) from baseline to 1, 2, and 3 months | 3 months
  Oxygen consumption and carbon dioxide production will be measured in a resting condition via indirect calorimetry (Quark RMR w/CPET, version 9.1) for 30 minutes.
Changes in respiratory quotient from baseline to 1, 2, and 3 months | 3 months
  Respiratory quotient variations will be measured in a resting condition via indirect calorimetry (Quark RMR w/CPET, version 9.1) for 3 hours. The first 30 minutes will be conducted in a fasting condition. After that, a blood collection will be taken to measure insulin concentration and the participants will consume a standardized meal (2 bottles of Boost Complete Nutritional Drink). After that, indirect calorimetry will be performed for 2 hours, with a blood collection every 60 minutes. This procedure will take place after an overnight fast of 10 hours and refraining from exercise and alcohol ingestion in the previous day.
Changes in metabolic flexibility from baseline to 1, 2, and 3 months | 3 months
  Oxygen consumption and carbon dioxide production will be measured in a resting condition via indirect calorimetry (Quark RMR w/CPET, version 9.1) for 2 hours and 30 minutes. The first 30 minutes will be conducted in a fasting condition. After that, a blood collection will be taken to measure insulin concentration and the participants will consume a standardized meal (2 bottles of Boost Complete Nutritional Drink). After that, indirect calorimetry will be performed for 2 hours, with a blood collection every 60 minutes. This procedure will take place after an overnight fast of 10 hours and refraining from exercise and alcohol ingestion in the previous day.
Changes in maximal aerobic capacity from baseline to 1, 2, and 3 months | 3 months
  To determine maximal aerobic capacity, a ramp incremental protocol to exhaustion will be performed on a cycle ergometer (Monark 839E). The assessment will start at 20 Watts/min and then the workloads will increase in increments of 5-20 Watts/min. Cadence: 60 rotations/min. All tests will be monitored using a 12-lead electrocardiogram and all data will be monitored and recorded using Omnia software. Expired and inspired gases are continuously analyzed, breath-by-breath, through a portable gas analyzer (Quark RMR w/CPET). Participants will exercise until at least one of the following objective test criteria is reached: (1) respiratory exchange ratio reached 1.1 or higher; (2) participants reached predicted maximal heart rate; and (3) oxygen uptake did not increase in spite of increasing workload. VO2peak will be defined as the highest 20 seconds value for peak oxygen consumption attained in the last minute.
Changes in peak power output (PPO) from baseline to 1, 2, and 3 months | 3 months
  The cardiopulmonary exercise test (CPET) will be used to assess each participant's PPO. To determine PPO, a ramp incremental protocol to exhaustion will be performed on a cycle ergometer (Monark 839E, Kroons Vag, Sweeden). Participants will start the assessment at 20 Watts/min and then the workloads will increase in increments of 5-20 Watts/min (according to personal cardiopulmonary response to exercise during the first minute), while on a constant pedal frequency of 60 rotations/min. All the tests will be monitored using a 12-lead electrocardiogram personal computer-based acquisition module and all data, including heart rate, will be monitored and recorded using Omnia software (Cosmed, Rome, Italy). During this test, expired and inspired gases are continuously analyzed, breath-by-breath, through a portable gas analyzer (Quark RMR w/CPET, version 9.1, Cosmed, Rome, Italy). PPO will be defined as the last ramp stage achieved by the participants during the incremental output.
Changes in glucose from baseline to 1, 2, and 3 months | 3 months
  Fasting blood samples will be collected at baseline and at the end of each of the 2-week exercise intervention blocks by APDP certified staff. Blood collection will be performed in a seated position from the antecubital vein, at rest, after an overnight fast, into dry tubes and into tubes containing ethylenediamine-tetraacetic acid, an anticoagulant. Biological samples will be centrifuged at 500 g at 4°C for 15 minutes and plasma samples will be frozen at -80 °C for posterior analysis. Blood samples will be delivered on ice to the APDP for glucose analysis. All samples will be used once for analysis and disposed of after following the APDP clinical protocols.
  From serum blood samples, glucose will be analyzed using colored enzymatic tests in an automated analyzer (auto analyzer Olympus AU640, Beckman Coulter).
Changes in insulin from baseline to 1, 2, and 3 months | 3 months
  Fasting blood samples will be collected at baseline and at the end of each of the 2-week exercise intervention blocks by APDP certified staff. Blood collection will be performed in a seated position from the antecubital vein, at rest, after an overnight fast, into dry tubes and into tubes containing ethylenediamine-tetraacetic acid, an anticoagulant. Biological samples will be centrifuged at 500 g at 4°C for 15 minutes and plasma samples will be frozen at -80 °C for posterior analysis. Blood samples will be delivered on ice to the APDP for insulin analysis. All samples will be used once for analysis and disposed of after following the APDP clinical protocols.
  Serum insulin will be analyzed using an electrochemiluminescence immunoassay (Liaison, Diasorin).
Changes in glucose (CGM) from baseline to 1, 2, and 3 months | 3 months
  24-hour blood glucose levels will be measured with a CGM monitor (CGM - iPro2 Professional Continuous Glucose Monitoring, MiniMed; Medtronic, Northridge, CA, USA) connected to a glucose sensor (Enlite Glucose Sensor MiniMed; Medtronic, Northridge, CA, USA). The sensor will be placed subcutaneously on the right side of the abdomen prior to eating any of the standardized pre-made meals with macronutrient distribution based on the recommended dietary guidelines (either breakfast, lunch, snack or dinner). The monitor will provide interstitial glucose values every 5 minutes and will be removed 24 hours later. During this 24-hour period, all meals will be standardized and provided to the participants. In addition, the time of all medications taken will be recorded.
Quantify the differences in the number of responders and low-responders for glycemic control and other health-related outcomes for individuals with T2DM and age-matched overweight/obese older adults. | 3 months
  To quantify responder variability to exercise at the different times of the day, the investigators will first calculate the technical error of the 24h AUC measurement provided by the CGM for each participant. This value will be calculated by taking the difference between the repeated baseline measures at each exercise block. The observed changes in AUC for each participant will be adjusted by the technical error for that participant. Individuals will be classified has having a true response to exercise at the given time of day if their adjusted change score is beyond the calculated minimal clinically important difference (MCID) (i.e., effect size of 0.2 x baseline between-subject SD). This technique for establishing responder thresholds has previously been suggested and used by others as a viable approach for assessing individual response variability.

CONTACTS AND LOCATIONS:
Overall Officials: João B Magalhães, PhD, Principal Investigator — Faculdade de Motricidade Humana - Universidade de Lisboa
Locations (1):
- Faculdade de Motricidade Humana, Cruz Quebrada, Oeiras, Portugal

REFERENCES:
- [Derived] Magalhaes JP, Oliveira EC, Hetherington-Rauth M, Jesus F, Rodrigues MC, Raposo JF, Ribeiro RT, Caetano C, Sardinha LB. The Ex-Timing trial: evaluating morning, afternoon, and evening exercise on the circadian clock in individuals with type 2 diabetes and overweight/obesity-a randomized crossover study protocol. Trials. 2024 Aug 6;25(1):526. doi: 10.1186/s13063-024-08335-y. PMID 39107793